CLINICAL TRIAL: NCT03974932
Title: A Phase 3b, Open-Label Study of HTX-011 as Part of a Scheduled Non-Opioid Multimodal Analgesic Regimen in Subjects Undergoing Total Knee Arthroplasty
Brief Title: Total Knee Arthroplasty (TKA) Study of HTX-011 in an Multimodal Analgesic Regimen (MMA) Regimen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Heron Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HTX-011-306
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Analgesia
Keywords: total knee arthroplasty; postoperative pain; multimodal analgesia
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Ibuprofen; Acetaminophen; Celecoxib; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- Cohort 1 (Experimental): HTX-011 + MMA
  Interventions: Drug: HTX-011; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Celecoxib; Device: Luer Lock Applicator
- Cohort 2 (Experimental): HTX-011 + MMA
  Interventions: Drug: HTX-011; Drug: Ibuprofen; Drug: Acetaminophen; Drug: Celecoxib; Device: Luer Lock Applicator
- Cohort 3 (Experimental): HTX-011 + MMA
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen; Drug: Celecoxib; Drug: +/- Bupivacaine HCl; Device: Luer Lock Applicator; Drug: HTX-011
- Cohort 4 (Experimental): HTX-011 + MMA
  Interventions: Drug: HTX-011; Drug: Ibuprofen; Drug: Acetaminophen; Device: Luer Lock Applicator

INTERVENTIONS:
Drug: HTX-011 — Dual-acting local anesthetic. Dose 1.
  Arms: Cohort 1; Cohort 2; Cohort 4
Drug: Ibuprofen — NSAID.
Drug: Acetaminophen — Analgesic.
Drug: Celecoxib — NSAID.
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: +/- Bupivacaine HCl — Local anesthetic.
  Arms: Cohort 3
Device: Luer Lock Applicator — Applicator for instillation.
Drug: HTX-011 — Dual-acting local anesthetic. Dose 2.
  Arms: Cohort 3

SUMMARY:
Phase 3b, open-label single-arm study in which all subjects receive HTX-011 as part of a scheduled non-opioid MMA regimen.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled to undergo primary unilateral TKA under spinal anesthesia.
* Has not previously undergone TKA in either knee.
* Has an American Society of Anesthesiologists (ASA) Physical Status of I, II, or III.
* Is able to walk at least 20 feet with optional use of a 4-legged walker for balance.
* Female subjects are eligible only if not pregnant, not lactating, not planning to become pregnant during the study, sterile; or is at least 2 years post-menopausal; or is in a monogamous relationship with a partner who is surgically sterile; or using acceptable contraceptives.

Exclusion Criteria:

* Has a planned concurrent surgical procedure.
* Has other pre-existing concurrent acute or chronic painful physical/restrictive condition expected to require analgesic treatment in the postoperative period for pain.
* Has a contraindication or a known or suspected history of hypersensitivity or clinically significant idiosyncratic reaction to required study medications.
* Using or expected to use Factor IX Complex or anti-inhibitor coagulant concentrates during the study.
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months.
* Has taken NSAIDs within 10 days prior to the scheduled surgery with the exception of subjects on low-dose (≤100 mg) daily acetylsalicylic acid for cardioprotection.
* Has taken opioids within 24 hours prior to the scheduled surgery (3 days for long-acting).
* Has been administered bupivacaine within 5 days prior to the scheduled surgery.
* Has been administered any local anesthetic within 72 hours prior to the scheduled surgery.
* Has initiated treatment with medications within 1 month prior to study drug administration that can impact pain control.
* Has been administered systemic steroids within 5 half-lives or 10 days prior to administration of study drug.
* Received an investigational product or device in a clinical trial within 30 days or within 5 elimination half lives.
* Has a known or suspected history of drug abuse, a positive drug screen on the day of surgery, or a recent history of alcohol abuse.
* Has a medical condition such that, in the opinion of the Investigator, participating in the study would pose a health risk to the subject or confound the postoperative assessments.
* Is currently undergoing treatment for hepatitis B, hepatitis C, or HIV.
* Has uncontrolled anxiety, psychiatric, or neurological disorder that, in the opinion of the Investigator, might interfere with study assessments.
* Has acquired defective color vision or acute gastrointestinal ulcers, either of which could interfere with scheduled study medications.
* Has any chronic neuromuscular deficit of either femoral nerve function or thigh musculature.
* Has any chronic condition or disease that would compromise neurological or vascular assessments.
* Had a malignancy in the last year, with the exception of nonmetastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Has undergone 3 or more surgeries within 12 months.
* Has a body mass index (BMI) >39 kg/m2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Helen Keller Hospital, Sheffield, Alabama
  - Phoenix Clinical Research, LLC, Tamarac, Florida
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - First Surgical Hospital, Bellaire, Texas
  - Plano Surgical Hospital, Plano, Texas
  - Endeavor Clinical Trials, LLC., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects in Cohort 1 and Cohort 2 received the same Assigned Intervention (ie, HTX-011 400 mg/12 mg + celecoxib-containing MMA regimen) and results are pooled for the purpose of this Results Section.
Groups:
- Cohort 1 and Cohort 2 (Pooled): HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg + celecoxib-containing MMA regimen.
- Cohort 3: Group A: HTX-011 (bupivacaine/meloxicam), 300 mg/9 mg + celecoxib-containing MMA regimen.
- Cohort 3: Group B: HTX-011 (bupivacaine/meloxicam), 300 mg/9 mg and 100 mg bupivacaine HCl + celecoxib-containing MMA regimen.
- Cohort 4: HTX-011 (bupivacaine/meloxicam), 400 mg/12 mg + ibuprofen-containing MMA regimen.
Period: Overall Study
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Started | 66 | 14 | 16 | 20
Completed | 66 | 14 | 16 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4 | Total
Number analyzed (Participants) | 66 | 14 | 16 | 20 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 6 | 6 | 7 | 54
  >=65 years | 31 | 8 | 10 | 13 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (9.64) | 62.4 (8.88) | 66.8 (9.81) | 69.0 (8.82) | 65.1 (9.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 4 | 12 | 12 | 65
  Male | 29 | 10 | 4 | 8 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 1 | 3 | 5 | 29
  Not Hispanic or Latino | 46 | 13 | 13 | 15 | 87
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — The 1 participant in Cohort 2 listed as 'Unknown or Not Reported' includes Puerto Rican.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 6 | 3 | 3 | 5 | 17
    White | 59 | 11 | 13 | 15 | 98
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 66 | 14 | 16 | 20 | 116

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve (AUC) of the Visual Analogue Scale (VAS).
Description: The Visual Analog Scale (VAS) consists of a straight 10-cm line that represents pain ranging from "no pain" to "pain as bad as it could be". Subjects were asked to mark their current pain level on the line.
Time Frame: 12 through 48 hours
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
pain intensity score*hr | 155.57 (95.651) | 185.27 (86.898) | 161.36 (86.627) | 126.59 (118.431)

2. Secondary Outcome: Mean AUC of VAS Scores.
Description: as for outcome 1
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
pain intensity score*hr | 277.03 (164.004) | 319.81 (158.746) | 276.87 (146.578) | 216.18 (206.164)

3. Secondary Outcome: Mean AUC of the NRS of Pain Intensity at Rest (NRS-R).
Description: Pain intensity scores are assessed using an 11-point Numeric Rating Scale (NRS) (0-10) where 0 represents "no pain" and 10 represents "worst pain". NRS scores are measured at rest.
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: pain intensity score*hr
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
pain intensity score*hr | 309.89 (155.289) | 355.20 (161.377) | 311.00 (136.714) | 245.00 (200.369)

4. Secondary Outcome: Percentage of Subjects With Severe Pain.
Description: Severe Pain defined as a VAS score ≥7.5 cm.
Time Frame: 24 hours, 48 hours, 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants
  24 Hours | 26 | 4 | 5 | 6
  48 Hours | 29 | 5 | 5 | 6
  72 Hours | 23 | 5 | 5 | 7

5. Secondary Outcome: Mean Total Postoperative Opioid Consumption (in IV Morphine Milligram Equivalents [MME]).
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: MME, morphine milligram equivalency
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
MME, morphine milligram equivalency | 26.40 (23.229) | 31.50 (24.907) | 23.40 (14.484) | 17.62 (22.167)

6. Secondary Outcome: Percentage of Subjects Who Are Opioid-free
Time Frame: 72 Hours to Day 11
Measure: Number; unit: participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
participants | 25 | 4 | 3 | 10

7. Secondary Outcome: Percentage of Subjects Who Are Opioid-free Through 72 Hours Who Remain Opioid-free Through Day 11.
Time Frame: 72 hours through Day 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants | 9 | 1 | 0 | 5

8. Secondary Outcome: Median Time to First Opioid Rescue Medication.
Time Frame: Through 72 hours
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Hours | 6.12 [4.27 to 8.25] | 5.63 [2.12 to 19.48] | 9.96 [4.18 to 15.90] | 12.76 [5.80 to 47.10]

9. Secondary Outcome: Percentage of Subjects Who do Not Receive an Opioid Prescription at Discharge.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants | 41 | 8 | 12 | 13

10. Secondary Outcome: Percentage of Subjects Who do Not Receive an Opioid Prescription Between Discharge and the Day 11 Visit.
Time Frame: 72 hours through Day 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants | 44 | 8 | 8 | 17

11. Secondary Outcome: Percentage of Subjects Achieving a Score of "Good" or Better (>1) Pain Control Based on Patient Global Assessment (PGA).
Description: Patient's Global Assessment (PGA) of pain control is a 4-point scale in which subjects rate how well their pain has been controlled (0 = Poor; 1 = Fair; 2 = Good; 3 = Excellent).
Time Frame: 24 hours, 48 hours, 72 hours, Day 11
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants
  24 Hours | 60 | 10 | 14 | 16
  48 Hours | 61 | 11 | 14 | 16
  72 Hours | 66 | 12 | 15 | 18
  Day 11 | 50 | 11 | 11 | 15

12. Secondary Outcome: Median Time to First Ambulation Postsurgery.
Time Frame: 72 hours
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Hours | 20.66 [18.48 to 23.43] | 23.20 [6.08 to 54.62] | 26.72 [24.37 to 29.60] | 20.58 [5.83 to 23.92]

13. Secondary Outcome: Percentage of Subjects Unable to Participate in Each Rehabilitation Session Because of Pain.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants | 23 | 1 | 2 | 3

14. Secondary Outcome: Percentage of Subjects Who First Achieve an MPADSS Score ≥9.
Description: Subjects were assessed for readiness for discharge using the Modified Post-Anesthesia Discharge Scoring System (MPADSS) that assesses 5 clinical variables: vital signs, ambulation, nausea/vomiting, pain, and surgical bleeding, each on a 3-point scale of 0, 1, or 2 with 0 being the worst score and 2 being the best score. Subjects with an MPADSS score of 9 or 10 were considered ready for discharge.
Time Frame: 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24, hours, 36 hours, 48 hours, 60 hours, 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants
  Through 2 Hours | 15 | 2 | 2 | 0
  Through 4 Hours | 16 | 3 | 2 | 3
  Through 6 Hours | 21 | 6 | 5 | 7
  Through 8 Hours | 29 | 6 | 8 | 8
  Through 12 Hours | 38 | 7 | 9 | 8
  Through 24 Hours | 45 | 8 | 11 | 15
  Through 36 Hours | 52 | 12 | 13 | 18
  Through 48 Hours | 57 | 12 | 13 | 19
  Through 60 Hours | 57 | 12 | 15 | 19
  Through 72 Hours | 59 | 13 | 15 | 19

15. Secondary Outcome: Percentage of Subjects Who Are Discharged Home vs to a Skilled Nursing Facility.
Description: Number Analyzed represents Subjects who were discharged home.
Time Frame: 72 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Participants | 61 | 10 | 16 | 20

16. Secondary Outcome: Mean Overall Benefit of Analgesia Score (OBAS).
Description: Subjects were questioned about their overall benefit of analgesia. Overall benefit of analgesia score (OBAS) assesses current pain at rest, vomiting, itching, sweating, freezing, dizziness, and overall satisfaction with postoperative pain during the previous 24 hours. To calculate the OBAS score, each of the subscale scores (0=minimum; 4=maximum) are summed for a combined OBAS score. Possible scores could range from 0 to 28 with a lower score indicating greater benefit.
Time Frame: 24 hours, 48 hours, 72 hours, Day 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Scores on a scale
  24 Hours | 6.5 (2.75) | 7.4 (6.36) | 7.6 (3.24) | 5.9 (3.45)
  48 Hours | 5.7 (2.76) | 4.9 (1.44) | 5.9 (2.89) | 5.3 (2.57)
  72 Hours | 5.1 (2.46) | 4.1 (1.77) | 4.9 (1.88) | 4.8 (2.29)
  Day 11 | 5.0 (2.43) | 5.2 (2.08) | 4.9 (2.08) | 4.9 (2.07)

17. Secondary Outcome: Mean Total TSQM-9 Score
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) contains 9 items assessing Effectiveness, Convenience, and Global Satisfaction domains. Responses to items are rated on a 5-point or 7-point rating scale. Scores for each domain are computed by adding the TSQM items in each domain and then transforming the values in to a composite score ranging from 0 to 100, with higher scores representing higher satisfaction.
Time Frame: 72 hours through Day 11
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 66 | 14 | 16 | 20
Scores on a scale
  Global Satisfaction Domain - 72 Hours | 86.9 (15.53) | 77.0 (22.62) | 89.3 (14.75) | 86.8 (13.57)
  Effectiveness Doman - 72 Hours | 86.4 (18.09) | 80.2 (20.52) | 84.0 (14.61) | 81.9 (15.39)
  Convenience Domain - 72 Hours | 90.1 (12.03) | 84.5 (17.18) | 93.1 (13.07) | 86.9 (16.45)
  Global Satisfaction Domain - Day 11 | 78.0 (22.39) | 74.5 (27.27) | 72.8 (21.22) | 82.9 (18.16)
  Effectiveness Doman - Day 11 | 76.3 (21.18) | 69.4 (29.13) | 69.4 (29.13) | 67.0 (24.80)
  Convenience Domain - Day 11 | 90.1 (12.03) | 86.9 (15.50) | 80.9 (15.31) | 90.6 (12.24)

18. Secondary Outcome: Maximum Concentration (Cmax)
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 65 | 14 | 16 | 20
ng/mL
  Bupivacaine | 566 (273) | 534 (175) | 742 (268) | 851 (288)
  Meloxicam | 238 (96.8) | 247 (89.0) | 251 (104) | 385 (161)

19. Secondary Outcome: Time of Occurrence of Maximum Concentration (Tmax)
Time Frame: 72 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
Number analyzed (Participants) | 65 | 14 | 16 | 20
hours
  Bupivacaine | 21.05 [1.07 to 49.83] | 20.54 [3.98 to 37.27] | 20.14 [2.10 to 37.02] | 22.48 [8.05 to 48.63]
  Meloxicam | 47.13 [18.38 to 49.83] | 58.58 [23.65 to 73.28] | 37.17 [20.35 to 71.43] | 48.58 [20.85 to 73.37]

ADVERSE EVENTS:
Time Frame: From the time the subject signed the informed consent form (ICF) through the Day 29 Visit.
Description: At each level of summarization (any event and Preferred Term), subjects reporting more than one adverse event are counted only once.
Arm/Group | Cohort 1 and Cohort 2 (Pooled) | Cohort 3: Group A | Cohort 3: Group B | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/14 | 0/16 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/66 | 0/14 | 0/16 | 2/20
Other Adverse Events (participants affected / at risk) | 56/66 | 12/14 | 14/16 | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and Cohort 2 (Pooled) (N=66) | Cohort 3: Group A (N=14) | Cohort 3: Group B (N=16) | Cohort 4 (N=20)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and Cohort 2 (Pooled) (N=66) | Cohort 3: Group A (N=14) | Cohort 3: Group B (N=16) | Cohort 4 (N=20)
Dizziness (Nervous system disorders) | 9 | 1 | 2 | 1
Headache (Nervous system disorders) | 2 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 3 | 3 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 3 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 33 | 6 | 11 | 6
Vomiting (Gastrointestinal disorders) | 17 | 3 | 7 | 5
Constipation (Gastrointestinal disorders) | 10 | 3 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 3 | 3 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 3 | 1 | 0
Peripheral swelling (General disorders) | 3 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 1 | 1
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 9 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Incision site oedema (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 4 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT03974932/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03974932/SAP_001.pdf